CLINICAL TRIAL: NCT05670457
Title: Diosmin as Adjuvant Therapy in Treatment of Non-bleeding Peptic Ulcer
Status: Unknown | Phase: Phase 3 | Type: Interventional
Last Known Status: Recruiting
Sponsor: Tanta University (Other)
Responsible Party: Principal Investigator, Ahmed Gamal Salah Abdelfatah, principal investigator, Tanta University
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: diosmin peptic ulcer
Record Dates: First submitted 2023-01-02; First posted 2023-01-04 (Actual); Last update posted 2023-01-04 (Actual); Status verified 2023-01

CONDITIONS: Non-bleeding Peptic Ulcer
MeSH Terms: interventions — Diosmin

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Control group (No Intervention): this group will include 22 patients who will receive anti peptic ulcer only for 2 months.
- Diosmin group (Active Comparator): this group will include 22 patients who will receive anti peptic ulcer and diosmin 500 mg twice daily for 2 months.
  Interventions: Drug: Diosmin

INTERVENTIONS:
Drug: Diosmin — diosmin 500 mg twice daily
  Arms: Diosmin group

SUMMARY:
The aim of the study is to evaluate the safety and efficacy of diosmin as adjuvant therapy in treatment of non-bleeding peptic ulcer patients.

ELIGIBILITY:
Inclusion Criteria:

-. Age 25-65 years old.

* Patients of both gender (male and female).
* Non-bleeding Peptic ulcer Patients (duodenal &gastric) diagnosed by endoscopy.

Exclusion Criteria:

* The presence of other factors that can lead to gastric bleeding other than peptic ulcer.

  * Patients with cancerous disease
  * Breast-feeding.
  * Surgically altered stomach ( bariatric surgery),
  * Patient with liver disease.
* Bleeding & perforated peptic ulcer.

Ages: 25 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 44 (Estimated)
Dates: Start 2022-06-30 (Actual); Primary Completion 2024-06 (Estimated); Study Completion 2025-06 (Estimated)

PRIMARY OUTCOMES:
assesment of improvement of symptoms as indicated by change in SAGIS scale. | 2 months
  patients will undergo clinical assessment according to SAGIS scale at baseline and 2 months

SECONDARY OUTCOMES:
change in Malondialdehyde (MDA) serum levels. | 2 months
  blood samples will be collected at baseline and 2 months.
change in Prostaglandin E2 (PGE2) serum levels. | 2 months.
  blood samples will be collected at baseline and 2 months.
change in Endothelin-1 (ET-1) serum levels. | 2 months
  blood samples will be collected at baseline and 2 months.
change in b-cell lymphoma 2(bcl-2) serum levels. | 2 months
  blood samples will be collected at baseline and 2 months.

CONTACTS AND LOCATIONS:
Locations (1):
- Tanta University, Tanta, El Gharbia, Egypt